CLINICAL TRIAL: NCT02602717
Title: The Evaluation of the Diagnostic Properties of Intra-operative In-situ Thyroglobin Levels of Cervical Lymph Nodes, in the Discrimination Between Benign and Malignant Lymph Nodes in Thyroid Cancer: a Prospective Multicentre Study.
Acronym: Tgcyto
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-06; RC12_3625 (Other: APHM)
Record Dates: First submitted 2015-10-22; First posted 2015-11-11 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Thyroid Cancer
Keywords: follicular origin
MeSH Terms: conditions — Thyroid Neoplasms

ARMS (1):
- thyroid cancer (Experimental)
  Interventions: Other: lymph nodes cyto-punction

INTERVENTIONS:
Other: lymph nodes cyto-punction

SUMMARY:
Cytological examination of punctured lymph nodes is the gold standard for confirming metastatic lymph node spread of differentiated thyroid cancers. In order to increase the diagnostic sensitivity of fine-needle cyto-punctured lymph nodes, an assessment of Tg levels of the aspirate could be included. Although this technique has been well proven, many uncertainties remain, especially with regards to a pathological cut-off value and its clinical utility when the thyroid is still intact. This uncertainty is mainly due to discordancy between low Tg levels found in cytopunctured lymph nodes with normal cytology, and their final histopathological analyses.

To eliminate this uncertainty, cyto-punction will be performed intra-operatively after localizing and isolating the target lymph nodes for assessment of cytology and Tg values. The thyroid gland might be present or absent (already operated) depending on the case. Finally, the cyto-punctured lymph nodes will be excised for complete histopathological analysis. In order to determine whether the Tg values are appropriate in cases where the thyroid is intact, a control group has been included (First operation for thyroid cancer or benign pathology). To eliminate the possible iatrogenic risks of lymph node dissection and resection in patients for whom it is not indicated, only lymph nodes found along the incision path for neuromonitoring of the recurrent laryngeal nerve (performed systematically) will be analysed and excised.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 years and above, male or female, with a valid social security coverage;
* Subject willing to participate in the study with a signed informed consent;
* Subject being operated for a papillary thyroid cancer, re-operated for persistent/relapsed lymphadenopathy, or for benign thyroid pathology (Graves disease, multinodular goitre, toxic nodule);
* Subject having had a blood test for plasma Tg levels and circulating anti-Tg antibodies in the week preceding the surgical intervention.

Exclusion Criteria:

- Subjects presenting with thyroid cancers of non follicular origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-02-18 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
thyroglobin levels dosage | 7 days

SECONDARY OUTCOMES:
Plasma Tg levels | 7 days
circulating anti-Tg antibodies levels | 7 days
Detection of tumor cells by staining with May-Grünwald Giemsa of lymph node cytology elements : | 15 days
Detection of tumors by lymph node histology | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — APHM
Locations (1):
- APHM, Marseille, France